CLINICAL TRIAL: NCT04452253
Title: Associations of Serum Total Antioxidant Capacity and Sleep or Psychiatric Symptoms in Employees Experiencing High Levels of Stress Before and After the Intake of Probiotics
Brief Title: Psychiatric Symptoms in Employees Experiencing High Levels of Stress Before and After the Intake of Probiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Collaborators: Bened Biomedical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shu-I Wu, Senior Attending Physician, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19CT013be
Record Dates: First submitted 2020-06-10; First posted 2020-06-30 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Probiotics

STUDY DESIGN:
Intervention Model Description: Sub-project 1 is a RCT study (Nurses) Sub-project 2 is an open label design (IT Employees)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PS128 (Experimental): The PS128, which belongs to Lactobacillus plantarum subsp. plantarum, 2 caps daily use and used in both sub-project 1 and 2.
  Sub-project 2 (Open label) for IT specialists only take PS128.
  Interventions: Dietary Supplement: PS128
- PS23 live (Experimental): The PS23 belongs to Lactobacillus paracasei group, 2 caps daily use, only used in sub-project 1.
  Interventions: Dietary Supplement: PS23 live
- PS23 heat-treated (Experimental): PS23 heat-treated, 2 caps daily use, only used in sub-project 1.
  Interventions: Dietary Supplement: PS23 heat-treated
- Placebo (Placebo Comparator): The placebo capsule contains microcrystalline cellulose, 2 caps daily use, only used in sub-project 1.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: PS128 — PS128 belongs to Lactobacillus plantarum subsp. plantarumand. Probiotic capsules contain 10 billion CFU (colony forming units) of PS128
  Arms: PS128
Dietary Supplement: PS23 live — PS23 belongs to Lactobacillus paracasei group.Probiotic capsules contain 10 billion CFU (colony forming units) of PS23
  Arms: PS23 live
Dietary Supplement: PS23 heat-treated — The PS23 heat-treated probiotic capsule contain 10 billion of PS23 cells.
  Arms: PS23 heat-treated
Other: Placebo — The placebo capsule contains microcrystalline cellulose.
  Arms: Placebo

SUMMARY:
Sub-project 1 Background:With the increasing number of shift workers required for social and economic activities, increasing prevalence of metabolic diseases has been found in this group of people. Although reasons for this include reduced physical activity owing to unfixed working hours, lack of sleep or disturbances in the circadian rhythm may also be related to the occurrences of type 2 diabetes or metabolic syndrome. The mechanism may be due to sleep deprivation induced activation of the hypothalamic- pituitary- adrenal axis (HPA axis) that affects blood glucose metabolism. The gut brain axis might adjust the HPA axis via the bottom-up pathway through vagus nerve, the neuroendocrine system, or the immune system. It is also possible that physiological or psychological stressors might influence intestinal function through the top-down pathways. Associations between microbiota and many chronic diseases, including metabolic syndrome, diabetes, obesity, neurodegenerative diseases, or mental diseases have been investigated in recent years. However, the application of using probiotics in treating sleep disorders is still lacking. The probiotics used in this proposal are selected to be more related to mental conditions. The PS128, which belongs to Lactobacillus plantarum subsp. plantarum and PS23 belongs to Lactobacillus paracasei group. Both PS128 and PS23 probiotic capsules contain 10 billion CFU (colony forming units) of PS128 or PS23. The PS23 heat-treated probiotic capsule contain 10 billion PS23 cells.

The main research hypothesis: Is it possible to develop the relevant probiotic treatment model?Our intended analysis was set a priori to analyze each probiotic vs. the placebo.

Sub-project 2 Information technology (IT) is an industry related to productions of computers, information processing, or telecommunications. Such industry highly relies on the knowledge and solutions provided by professional IT specialists. Literature has described that the subjective stress scores were higher in IT specialists that developed diabetes, hypertension, and depression. Specific probiotics, also known as psychobiotics, may have the effects of alleviating levels of stress and mood symptoms. Therefore this open-label designed, single arm, baseline-controlled trial aiming to examine whether an 8-week intervention of a novel psychobiotic Lactobacillus plantarum PS128TM (PS128TM), may improve self-perceived stress and mood symptoms among high-stress IT specialists.

DETAILED DESCRIPTION:
Sub-project 1 Materials

1. Probiotics The probiotics used in this proposal are selected to be more related to mental conditions. The PS128, which belongs to Lactobacillus plantarum subsp. plantarum. Administration of probiotics for 4 weeks in animal experiments showed significant improvements in depression and anxiety behaviors, and increased mobility in mice (Liu et al., 2016). The concentration of dopamine in the prefrontal cortex, which was reduced due to depression, was also restored by feeding PS128 (Liu et al., 2016). PS23 belongs to Lactobacillus paracasei group. In animal experiments, both live and heat-treated bacteria have the effect of improving depression and anxiety behaviors. The strains used in this study are food usable bacteria listed on the front of the Food and Drug Administration in Taiwan. The products have been sold in Taiwan in 2015 and there have been no serious adverse reactions. Relevant clinical studies have been reviewed by Institutional Review Boards in multiple hospitals (including the National Taiwan University Children's Hospital, Kaohsiung Kai-Syuan Psychiatric Hospital, Wanfang Hospital, Antai Hospital, and National Yangming University). These probiotics and placebo will be provided by the Yifu Biomedical Company Ltd. The probiotic powder contains no lactose and can be eaten by people with lactose intolerance. The placebo capsule contains microcrystalline cellulose. Both PS128 and PS23 probiotic capsules contain 10 billion CFU (colony forming units) of PS128 or PS23. The PS23 heat-treated probiotic capsule contain 10 billion PS23 cells. These products should be stored in the refrigerator and be protected from light. The probiotics and placebo used in the study are all edible fungi or food supplements approved by the Food and Drug Administration. There are no data on serious potential risks or side effects. Only a few gastric discomfort such as bloating or diarrhea have been reported.

Monitoring of adverse events and adverse reactions includes soft stools, flatulence, or diarrhea will be used for safety and tolerability assessment.

A total of 2 assessments and blood draws (week 0 and 8+1 weeks) will be required during the study period. Subjects will be invited to participate in the study (V0) and a questionnaire will be assessed. Those who meet the inclusion criteria will be assessed for baseline (V1), and the app for working hours recording and Rhythm (mobile phone schedule) must be installed to participants' mobile phones to record the working hours in the hospital. The once daily test capsules will be consumed the next day after the evaluation for 8 weeks until week 8 +1 (V2). At V2, a second assessment will be performed. The time of the second assessment needs to be the same as the first assessment. For example, the first assessment is for the day shift, and the second assessment must be for the day shift. The number of days consumed by each subject may be inconsistent, at least 28 days, and up to 35 days. Subjects are required to provide a working schedule for the study period for the second assessment to allow the investigator to match the assessment results for the analysis.

Research methods:

1. Investigators will enroll 240 nursing, psychologists and social workers who are working in the chronic and acute wards to participate. Participants will be evaluated in overall physical and mental health, sleep disturbances. 60 electronic employees will also be enrolled, participants will be evaluated in overall physical and mental health, sleep disturbances.
2. Blood TAC, Cortisol and DHEAS will be examined before and after administration of probiotics and placebo.
3. Subjects will need to complete several self-test scales, including the Questionnaire (PHQ-9), State-trait Active Inventory (form YA), Insomnia Severity Index (ISI), Buss Perry Offensive Scale, Quality of Life and Satisfaction Survey, 10 cm Visual Analogue Scale for Gastrointestinal Symptom and stress, Profile of Mood States (POMS) and Computerized Selective Attention Test.
4. In this study, double blind design will be adopted for subproject one and open label design will be adopted for subproject two. After consenting, participants will complete the above baseline assessment. All participants will then be randomly assigned to probiotic or placebo groups according to a computer-generated random number table. These two groups will be administered with probiotics or placebo for 8 weeks.

For the sub-project 2, all the participants will complete the baseline assessment and administered with probiotics for 8 weeks.

Statistics

1. General Considerations Data will be entered and error-checked by the Project Coordinator on IBM-compatible/Macintosh computers present both in the Psychological & Behavioral Science Research Laboratory in Mackay Memorial Hospital. The process of data entry, including preparation of data harvesting forms, database fields, data entry, and checking by editors will be supervised by the staff of the Psychological & Behavioral Science Research Laboratory, with extensive experience in both clinical trials and longitudinal studies with large data sets. Once the data set is entered and checked, analyses will be conducted using SPSS software. An "intent to treat" analysis examining all patients randomized to the trial will be performed to preserve the effect of randomization.
2. Power determination for the test of null hypothesis The power analysis will be conducted using the effect size from previous publications and the relevant studies of probiotics intervention. A minimally significant difference in PSS or ISI changes between treatments would be defined as a reduction of 20% or more in the score levels. Based on a power of 80% and assuming a 30% dropout rate and an alpha level of 0.05, a sample of 500 participants (120 per group) will be required. All results will be analyzed using an intent-to-treat analysisbased on treatment assignment, whether they complete treatment or not. It will also conduct a per-protocol analysis based on 'treated' participants, defined as those who received treatment and completed assessments at 0 and 8+1 weeks after allocation. To test the adequacy of randomization, it will conduct between group comparisons of baseline characteristics on all measures, using t tests for continuous variables and chi-square tests for dichotomous variables. Two tailed P-values<0.05 is considered significant. All analyses will be performed with SPSS version 12.0. To define better the link between changes in questionnaires and treatment response, changes in assessment scores will be assessed within the following categories according to treatment response as stated in previous literature: for PSS, ISI, STAI: 0% improvement; >0 to <=10% improvement; >10 to <=20% improvement and >20% improvement. Finally, to ensure that the observed effect will not better explained by changes in medication during follow-up or by antidepressant treatment, these two variables (changes in medication yes/no and taking antidepressant yes/no) will also be added into the models as covariates. The results of regression models will be presented as standardized regression coefficients (b) with 95% confidence intervals that can be interpreted as effect size. The threshold of significance was P=0.05.

For the sub-project 1 our intended analysis was set a priori to analyze each probiotic vs. the placebo.

Potential Benefits:

To the patients:

It may be possible to improve the stress, sleep or gastrointestinal symptoms of high-pressure nurses by supplementing probiotics.

To the participating researchers:

All participating assessors will be able to master the interview skills after the intensive interviewer training, in particular, familiar with semi-structured psychiatric interview and a package of self-report questionnaires. The laboratory researcher will be able to master the laboratory skills of performing epigenetic analysis, which can also be helpful in extending his research experience.

Scientific expectations:

The study will fill the research gap of shift work, metabolism, and probiotics in generally healthy high stress nursing staff. The results will provide empirical evidence for Asian scientists where there is still a lack of studies linked to changes before and after protiotics intervention. The knowledge for probiotics towards health promotion is expected to be increase and hope to lead to more personalized stratification for disease-risk models and for targeting effective interventions.

Sub-project 2 Materials: Probiotics The probiotics used in this proposal are selected to be more related to mental conditions. The PS128, which belongs to Lactobacillus plantarum subsp. plantarum.

Method:

IT specialists from a large IT company in Northern Taiwan were invited and first screened by the Perceived Stress Scale (PSS) 10 items version. Participants with a PSS-10 items score of 27 or higher were included in our study. Those currently under antibiotic or psychotropic treatments, have cancer, or other chronic physical or mental diseases were excluded. Two capsule that contained 300 mg of PS128TM powder, equivalent to 10 billion colony forming units, were suggested to be taken daily by the included participants. Other self-report measures included the Job Stress Scale, Visual Analogue Scale of Stress, the Insomnia Severity Index, the State and Trait Anxiety Index, The Questionnaire for Emotional Trait and State, the Patient Health Questionnaire, the Quality of Life Enjoyment and Satisfaction Questionnaire, and the Gastrointestinal Severity Index. Objective measures included Saliva levels of stress biomarkers include cortisol, α-amylase, Immunoglobulin A (IgA), lactoferrin, and lysozymes, and Tests on Attentional Performance.

ELIGIBILITY:
Sub-project 1

Inclusion Criteria:

* Full-time nursing staff from Mackay Memorial Hospital, including wards and special units.
* Age 20 to 60 years old.
* Perceived Stress Scale (PSS) 10- questions version, with a cutoff point of 27 points or more.

Exclusion Criteria:

* Have taken or are receiving antibiotics within one month.
* Probiotics used in powder, capsule or tablet in two weeks (except for Yogurt, Yogurt, Yakult and other related foods)
* Patients with hepatobiliary gastrointestinal tract who have undergone surgery
* Patients with past or present inflammatory bowel disease
* Those with a history of cancer
* Those who are allergic to lactic acid bacteria
* Currently taking medication to treat acute or chronic diseases or sleep disorders

Sub-project 2

Inclusion Criteria:

* Age 20 to 60 years old.
* Perceived Stress Scale (PSS) 10- questions version, with a cutoff point of 27 points or more
* Full time employee

Exclusion Criteria:

* Have taken or are receiving antibiotics within one month.
* Probiotics used in powder, capsule or tablet in two weeks (except for Yogurt, Yogurt, Yakult and other related foods)
* Patients with hepatobiliary gastrointestinal tract who have undergone surgery
* Patients with past or present inflammatory bowel disease
* Those with a history of cancer
* Those who are allergic to lactic acid bacteria
* Currently taking medication to treat acute or chronic diseases or sleep disorders

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Stress Scale (PSS) Score From Baseline to Change in Perceived Stress Scale (PSS) From Baseline to Week 12 Assessed for both sub-projects | From Baseline to 8 Weeks Assessed
  The PSS scores is a rating tool used to gauge the course of stree. The minimum total score possible is 0 and the maximum total score possible is 40. Higher values represent a worse outcome.

SECONDARY OUTCOMES:
Differences in the Job Stress Scale from the Ministry of Labor before and after consumption of probiotics. | From Baseline to 8 Weeks Assessed
  The job stress scale from Ministry of Labor is a rating tool used to gauge of stress.
Differences in Insomnia Severity index (ISI) before and after consumption of probiotics for both sub-projects. | From Baseline to 8 Weeks Assessed
  The ISI is a rating tool used to gauge of sleeping. Higher values represent a worse outcome.
Differences in the State and Trait Anxiety Index (STAI) before and after the consumption of probiotics for both sub-projects. | From Baseline to 8 Weeks Assessed
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.
Differences in the The Profile of Mood States (POMS) before and after probiotics consumption for both sub-projects‧ | From Baseline to 8 Weeks Assessed
  The Profile of Mood States (POMS) is a psychological rating scale used to assess transient, distinct mood states.
Changes in blood TAC (Total Antioxidant Capacity) before and after consumption of probiotics for sub-project 1. | From Baseline to 8 Weeks Assessed
  TAC is the biomarker for Oxidative stress
Changes in blood DHEA-S (Dehydroepiandrosterone sulfate) before and after consumption of probiotics for sub-project 1. | From Baseline to 8 Weeks Assessed
  DHEA-S (Dehydroepiandrosterone sulfate) is the biomarker for anti-aging，among the neuroactive steroids, dehydroepiandrosterone (3b-hydroxyandrost-5-ene-17-one, [DHEA]) and its sulfated metabolite DHEA sulfate (DHEAS) have been shown to be potent modulators of neural function, including neurogenesis, neuronal growth and differentiation, and neuroprotection. Highlighting the potential health significance of DHEA and DHEAS in humans, serum concentrations decrease steadily with age, with lowest concentrations present at the time many diseases of aging and neurodegeneration become apparent.
Changes in blood Cortisol before and after consumption of probiotics for sub-project 1 . Changes in saliva Cortisol before and after consumption of probiotics for sub-project 2 . | From Baseline to 8 Weeks Assessed
  Cortisol is a steroid hormone that is produced by the adrenal glands which sit on top of each kidney. When released into the bloodstream, cortisol can act on many different parts of the body and can help:
  body respond to stress or danger increase your body's metabolism of glucose control your blood pressure reduce inflammation. Cortisol is also needed for the fight or flight response which is a healthy, natural response to perceived threats. The amount of cortisol produced is highly regulated by your body to ensure the balance is correct.
Changes in blood High sensitivity CRP (hs CRP) before and after consumption of probiotics for sub-project 1. | From Baseline to 8 Weeks Assessed
  High-sensitivity C-reactive protein (hsCRP) is a marker of inflammation that predicts incident myocardial infarction, stroke, peripheral arterial disease, and sudden cardiac death among healthy individuals with no history of cardiovascular disease, and recurrent events and death in patients with acute or stable coronary syndromes.
Changes in saliva α-Amylase before and after consumption of probiotics for sub-project 2. | From Baseline to 8 Weeks Assessed
  Salivary alpha-amylase activity (sAA) is often considered to be surrogate markers of sympathetic activation in response to stress.
Changes in saliva Saliva IgA before and after consumption of probiotics for sub-project 2. | From Baseline to 8 Weeks Assessed
  Secretory IgA in saliva stands in a negative correlation to the level of the experienced stress
Changes in saliva lactoferrin before and after consumption of probiotics for sub-project 2. | From Baseline to 8 Weeks Assessed
  lactoferrin's multiple activities lie in its capacity to bind iron and to interact with the molecular and cellular components of hosts and pathogens. it can bind and sequester lipopolysaccharides, thus preventing pro-inflammatory pathway activation, sepsis and tissue damages.
Changes in saliva lysozyme before and after consumption of probiotics for sub-project 1. | From Baseline to 8 Weeks Assessed
  Lysozyme plays a pivotal role in the prevention of bacterial infections by attacking peptidoglycan in the bacterial cell wall.
Differences in times of deep and light sleep before and after consumption of probiotics for sub-projects 1. | From one week before Baseline to 8 Weeks Assessed
  Fitbit Charge 3 continuously tracks a variety of stats whenever subjects wear it. Data automatically syncs when in range of the Fitbit app throughout the day.
Differences in Trail making test before and after consumption of probiotics for sub-projects 1. | From Baseline to 8 Weeks Assessed
  The Trail Making Test is a neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy.[1] The test can provide information about visual search speed, scanning, speed of processing, mental flexibility, as well as executive functioning.
Differences in Insomnia Severity Index, ISI before and after consumption of probiotics | From Baseline to 8 Weeks Assessed
  The Insomnia Severity Index (ISI) is a brief instrument that was designed to assess the severity of both nighttime and daytime components of insomnia.
The Quality of Life, Enjoyment, and Satisfaction Questionnaire-16, QLESQ-16 | From Baseline to 8 Weeks Assessed
  The Quality of Life, Enjoyment, and Satisfaction Questionnaire-16 (QLESQ-16) is a valid, reliable self-report instrument for assessing quality of life.
Visual Analogue Scale-GI (VAS-GI) | From Baseline to 8 Weeks Assessed
  Visual Analogue Scale (VAS) consists of a line, 10 cm in length. Individuals point to or mark a spot on the line where they feel indicates their current their emotion, fatigue level and sleep quality. The score of emotion level is from 0cm (very nervous) to 10 cm (very relaxing). The score of fatigue level is from 0 cm (very energetic) to 10 cm (very sleepy). The score of sleep quality is from 0 cm (poor) to 10 cm (sleep well). The maximum total score is 100% (equal 10cm).

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Chieh Tsai, Ph.D, Study Director — Bened Biomedical Co., Ltd.
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Wu SI, Wu CC, Cheng LH, Noble SW, Liu CJ, Lee YH, Lin CJ, Hsu CC, Chen WL, Tsai PJ, Kuo PH, Tsai YC. Psychobiotic supplementation of HK-PS23 improves anxiety in highly stressed clinical nurses: a double-blind randomized placebo-controlled study. Food Funct. 2022 Aug 30;13(17):8907-8919. doi: 10.1039/d2fo01156e. PMID 35924970
- [Derived] Wu SI, Wu CC, Tsai PJ, Cheng LH, Hsu CC, Shan IK, Chan PY, Lin TW, Ko CJ, Chen WL, Tsai YC. Psychobiotic Supplementation of PS128TM Improves Stress, Anxiety, and Insomnia in Highly Stressed Information Technology Specialists: A Pilot Study. Front Nutr. 2021 Mar 26;8:614105. doi: 10.3389/fnut.2021.614105. eCollection 2021. PMID 33842519